CLINICAL TRIAL: NCT06022744
Title: An Exploratory Clinical Trial Evaluating LX109 Gene Therapy in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: An Exploratory Clinical Trial Evaluating LX109 Gene Therapy in Patients With nAMD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaodong Sun, Assessor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHGH-LX109
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: To Evaluate the Safety and Tolerability of Intravitreal Injection of LX109 in Patients With nAMD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LX109 (Experimental)
  Interventions: Drug: LX109

INTERVENTIONS:
Drug: LX109 — LX109 gene injection Specification: 0.2ml/bottle, 1.4×1012VG/ml Administration route: intravitreal injection, injection volume 0.05ml/eye

SUMMARY:
To evaluate the safety and tolerability of intravitreal injection of LX109 in patients with nAMD.

DETAILED DESCRIPTION:
In this study, 9 to 12 participants were enrolled in an open monocular, single dose escalation study design. Two dose groups were set up: low dose group (7×109 VG/ eye, 0.05ml) and high dose group (3.5×1010 VG/ eye, 0.05ml). Among them, 3 to 6 subjects were enrolled in low-dose group and 6 subjects were enrolled in high-dose group.

ELIGIBILITY:
Inclusion Criteria:

* 1) Informed consent must be signed before all assessments; 2) Male or female patients ≥50 years of age; 3) To investigate the presence of active CNV secondary to nAMD (occult or micromenorrhea) in the eye 4) When studying the baseline of the eye, use the ETDRS eye chart to test the BCVA of 19 to 73 letters (approximately equivalent to decimal notation) Recorded visual acuity 0.05-0.5); 5) Study eyes received at least 2 anti-VEGF treatments within 6 months. Note: For all subjects, only one eye was used as the "study eye" (i.e. the study eye receiving treatment). If both eyes of the subject meet the inclusion criteria, the eye with poor baseline vision will be selected as the study eye, or the eye with better vision may be selected for medical reasons or ethical requirements.

Exclusion Criteria:

* 1. In the investigator's judgment, concomitant eye diseases of the study eye at screening or baseline may cause subjects to fail to respond to study therapy or confuse the interpretation of study findings. For example, diabetic retinopathy, retinal vein obstruction, retinal retinal detachment, macular hiatus (stage 3 or 4), uveitis, vitreous macular traction affecting central vision, macular anterior membrane involving macular fovea or damaging macular structure, equivalent spherical lens ≤-8.00D of the study eye, etc.

  2. To investigate the presence of subretinal hyperreflective substance (SHRM) involving the fovea except CNV lesions; 3. Central serous chorioretinopathy (CSC) was confirmed in the study eyes at any time; 4. Study retinal detachment in the eye at any time; 5. Non-study eye BCV A less than decimal recorded visual acuity 0.05(<19 ETDRS letters); 6. The presence of uncontrolled glaucoma (defined as intraocular pressure ≥25mmHg after standard treatment) in the study eye; 7. Active intraocular or periocular inflammation or infection in the study eye or non-study eye; 8. To investigate the presence of CNV or macular edema secondary to causes other than AMD; 9. In the study, the refractive medium of the eye is seriously cloudy or the pupil cannot be sufficiently dilated, affecting BCVA or causing insufficient acquisition Clear eye imaging data, such as OCT, FFA, and fundus photography, affect researchers' observation of safety and efficacy.

Eye Treatment： 10. Internal eye surgery, such as vitrectomy, cataract phacoemulsification, trabeculectomy, or other filtering surgery, was performed within 3 months prior to baseline screening or study eye screening; 11. Study eyes screened or treated with intravitreal drug injections or drug-containing intraocular implants other than anti-VEGF drugs, such as intraocular corticosteroids, within 6 months prior to baseline; 12. Research eye or systemic have received gene therapy; 13. Study eyes screened or treated with macular laser photocoagulation or photodynamic therapy (PDT) or full vision membrane laser photocoagulation within 3 months prior to baseline; 14. Study eyes were screened or underwent YAG laser posterior capsulectomy or laser trabeculectomy or laser periiridectomy within 1 month prior to baseline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 4 weeks

SECONDARY OUTCOMES:
Change of mean BCVA score on the ETDRS visual acuity scale from baseline. | 4 weeks、24 weeks、52 weeks
  Changes of BCVA scores on the ETDRS visual acuity chart of the study eye from baseline at 4, 24 and 52 weeks after treatment with LX109.
Changes in mean eye CST from baseline at 4, 24 and 52 weeks after LX109 treatment were studied. | 4 weeks、24 weeks、52 weeks
The time after LX109 treatment to the first salvage treatment. | 52 weeks
Proportion of subjects receiving salvage treatment in the study eye at 24 weeks and 52 weeks after treatment with LX109. | 24 weeks、52 weeks
The number of times the eye received salvage treatment at 24 weeks and 52 weeks after treatment with LX109 was studied. | 24 weeks、52 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong WL, Su X, Li X, Cheung CM, Klein R, Cheng CY, Wong TY. Global prevalence of age-related macular degeneration and disease burden projection for 2020 and 2040: a systematic review and meta-analysis. Lancet Glob Health. 2014 Feb;2(2):e106-16. doi: 10.1016/S2214-109X(13)70145-1. Epub 2014 Jan 3. PMID 25104651
- [Background] Yang K, Liang YB, Gao LQ, Peng Y, Shen R, Duan XR, Friedman DS, Sun LP, Mitchell P, Wang NL, Wong TY, Wang JJ. Prevalence of age-related macular degeneration in a rural Chinese population: the Handan Eye Study. Ophthalmology. 2011 Jul;118(7):1395-401. doi: 10.1016/j.ophtha.2010.12.030. Epub 2011 Mar 27. PMID 21444116
- [Background] Ye H, Zhang Q, Liu X, Cai X, Yu W, Yu S, Wang T, Lu W, Li X, Jin H, Hu Y, Kang X, Zhao P. Prevalence of age-related macular degeneration in an elderly urban chinese population in China: the Jiangning Eye Study. Invest Ophthalmol Vis Sci. 2014 Sep 4;55(10):6374-80. doi: 10.1167/iovs.14-14899. PMID 25190650
- [Background] van Lookeren Campagne M, LeCouter J, Yaspan BL, Ye W. Mechanisms of age-related macular degeneration and therapeutic opportunities. J Pathol. 2014 Jan;232(2):151-64. doi: 10.1002/path.4266. PMID 24105633
- [Background] Mitchell P, Liew G, Gopinath B, Wong TY. Age-related macular degeneration. Lancet. 2018 Sep 29;392(10153):1147-1159. doi: 10.1016/S0140-6736(18)31550-2. PMID 30303083
- [Background] Khandhadia S, Cherry J, Lotery AJ. Age-related macular degeneration. Adv Exp Med Biol. 2012;724:15-36. doi: 10.1007/978-1-4614-0653-2_2. PMID 22411231
- [Background] Fleckenstein M, Keenan TDL, Guymer RH, Chakravarthy U, Schmitz-Valckenberg S, Klaver CC, Wong WT, Chew EY. Age-related macular degeneration. Nat Rev Dis Primers. 2021 May 6;7(1):31. doi: 10.1038/s41572-021-00265-2. PMID 33958600
- [Background] Holz FG, Tadayoni R, Beatty S, Berger A, Cereda MG, Cortez R, Hoyng CB, Hykin P, Staurenghi G, Heldner S, Bogumil T, Heah T, Sivaprasad S. Multi-country real-life experience of anti-vascular endothelial growth factor therapy for wet age-related macular degeneration. Br J Ophthalmol. 2015 Feb;99(2):220-6. doi: 10.1136/bjophthalmol-2014-305327. Epub 2014 Sep 5. PMID 25193672
- [Background] Cabral T, Lima LH, Mello LGM, Polido J, Correa EP, Oshima A, Duong J, Serracarbassa P, Regatieri CV, Mahajan VB, Belfort R Jr. Bevacizumab Injection in Patients with Neovascular Age-Related Macular Degeneration Increases Angiogenic Biomarkers. Ophthalmol Retina. 2018 Jan;2(1):31-37. doi: 10.1016/j.oret.2017.04.004. PMID 29376143